CLINICAL TRIAL: NCT03088592
Title: Electrophysiological Recordings of Deep Brain Stimulation in the Basal Ganglia
Acronym: DBSMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Markey Olson, Research Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHX-16-0017-70-06
Record Dates: First submitted 2017-03-02; First posted 2017-03-23 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Deep Brain Stimulation (Other): After informed consent is obtained, the patients will undergo routine DBS pre-operative evaluation and diagnostic testing. This includes a pre-operative 3T-MRI with and without gadolinium as well as pre-operative medical clearance by the patient's PCP or general practitioner and/or other medical specialist if necessary. They will also receive a baseline clinical evaluation including both motor function (Unified Parkinson's Disease Rating Scale on and off anti-parkinsonian medication) quality of life assessment (Parkinson's disease Questionnaire-39) and a full neuropsychological evaluation, if not already completed as part of the routine DBS candidacy evaluation within 2 months of surgery. Subjects will have medical clearance from their specialists and be be evaluated by an internal medicine physician prior to surgery and cleared to proceed.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Subjects will have awake or asleep DBS surgery with STN or GPi placement. Microelectrode recordings will define the electrophysiological target prior to lead implantation. Cortical recordings will be done using µECoG grids (2.0 x 0.8 cm) placed over the cortex through the same burr hole used for lead implantation. Neural recordings will be made continuously throughout the procedure: before, during, and after DBS, and at all levels of anesthesia. A pulse generator will be connected and implanted either during the operation or within 7-10 days post-operatively. Subjects will be admitted overnight for observation with anticipated discharge the next morning. The researchers will also be collecting other routine data points (length of surgery, stereotactic accuracy, length of hospital stay, and post-operative complications).
  Other Names: Activa PC Neurostimulator Model 37601 (Medtronic)

SUMMARY:
The pathology of Parkinson's disease (PD) and the mechanism of Deep Brain Stimulation surgery (DBS) are not completely understood. The recording data that is used routinely as part of the procedure to map the target structures, however, may be analyzed in order to better understand the neural network dynamics in PD. The purpose of the study is to perform simultaneous neural recordings from sub-cortical structures (e.g. subthalamic nucleus [STN] or globus pallidus internus [GPi]) and the cerebral cortex. These simultaneous recordings may provide insight in the pathology of PD and the mechanism of DBS. The researchers will also study the effects of anesthesia level on neuron synchronization . Recordings with micro-ECoG grid electrodes in the cortex show improved spatial resolution and these will be used to gain better understanding of cortical network dynamics and the synchronization with subcortical structures.

DETAILED DESCRIPTION:
Subjects will be identified exclusively from the researchers' clinical practice for evaluation of DBS surgical candidacy for Parkinson's disease. Once it is determined that a patient is an appropriate candidate for DBS placement (multidisciplinary team consensus) and has met inclusion criteria,the researchers will discuss the study with the subject and explain the rationale for the study as well as the implications the subject's participation has to their treatment. Informed consent will be obtained prior to study procedures being performed. Subjects will be in the study from the time of enrollment before surgery until all post-operative visits and tests are completed, usually by 6 months after surgery. Follow-up during this time will consist of the standard follow-up schedule that all patients who undergo DBS follow. This includes a clinic visit at 10-14 days, 12 weeks, and 6 months after DBS surgery. Subjects will also have a follow-up neurocognitive evaluation consisting of the same evaluative tests administered pre-operatively. These post-operative visits are standard for all patients undergoing DBS for Parkinson's.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease per Queens Square criteria
* Appropriate DBS candidate for multi-disciplinary team consensus
* Age 18 - 85 years of age
* Motor skills allowing for capability to complete evaluations
* Medically cleared for undergoing anesthesia and DBS surgery

Exclusion Criteria:

* Dementia per DSM-V criteria
* Medical or other condition precluding MRI
* History of supraspinal CNS disease other than PD
* Alcohol use of more than 4 drinks per day
* Pregnancy
* History of suicide attempt
* Currently uncontrolled clinically significant depression (BDI>20)
* History of schizophrenia, delusions, or currently uncontrolled visual hallucinations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Neural Recordings | pre-operative; intra-operative ; 10-14 post-operative; 12 week post-operative; 6 months post-operative
  Simultaneous neural recordings from sub-cortical structures (e.g. subthalamic nucleus [STN] or globus pallidus internus [GPi]) and the cerebral cortex will be collected. Recordings include action potentials and local field potentials from sub-cortical structures while subdural microelectrocorticography grids will be used to record local field potential from the cerebral cortex. Time, frequency, and phase relationships between action potentials and local field potentials will also be studied in the context of the level of anesthesia. Analysis of these simultaneous recordings, including assessing any changes, may provide insight in the pathology of PD and the mechanism of DBS.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — Barrow Brain and Spine physician with SJHMC privileges
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No